CLINICAL TRIAL: NCT07342608
Title: Safety and Performances of the LINEA Cardiac Pacing Lead Optimized for the Implantation in Interventricular Septum
Acronym: STARLIGHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLAI01 - STARLIGHT
Record Dates: First submitted 2025-11-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Bradycardia; Left Bundle Branch Area Pacing; Left Bundle Branch Pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LINEA cardiac pacing lead (Experimental)
  Interventions: Device: Use of LINEA cardiac pacing lead and FLEXIGO delivery catheter

INTERVENTIONS:
Device: Use of LINEA cardiac pacing lead and FLEXIGO delivery catheter — Use of LINEA cardiac pacing lead and FLEXIGO delivery catheter for implantation of pacemaker

SUMMARY:
The purpose of the clinical investigation is to evaluate the safety and performances of the new LINEA cardiac pacing lead, intended for placement at the interventricular septum.

ELIGIBILITY:
Inclusion criteria (phase I and II):

* Patient indicated for cardiac pacing according to the most recent guidelines from the European Society of Cardiology (ESC)
* Patient planned for a de novo implantation of an ALIZEA, BOREA or CELEA Single Chamber (SR) or Dual Chamber (DR) pacemaker from MicroPort CRM
* Patient planned for a catheter-guided ventricular pacing lead implantation in the interventricular septum area
* Patient's pacemaker with the remote monitoring functions accepted by the patient and planned to be activated

Exclusion criteria (phase I and II):

* Patient planned for a device upgrade, or a device or a lead replacement
* Patient with a congenital heart disease, hypertrophic cardiomyopathy or infiltrative cardiomyopathy
* Patient with a Left Ventricular Ejection Fraction (LVEF) ≤ 35%
* Patient already enrolled in another clinical investigation that could confound the results of this clinical investigation (e.g., clinical investigations involving intra-cardiac device)
* Patient having a contraindication for cardiac pacing system implantation (i.e. patient implanted with a defibrillator, patient for whom a single dose of steroid eluted by the pacing lead (e.g., dexamethasone sodium phosphate) is contraindicated, patient implanted with a tricuspid replacement heart valve, with prior tricuspid valve intervention or with a significant tricuspid valve disease that may lead to future replacement heart valve surgery)
* Patient with a life expectancy of less than 2 years
* Minor age patient (i.e. under 18 years of age)
* Incapacitated patient, under guardianship, kept in detention, refusing to cooperate or not able to understand the purpose of this clinical investigation
* Non-menopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
LINEA lead complication free rate at 3 months | 3 months after implantation
  Proportion of patients free from complication related to the LINEA lead. A complication is defined as a SADE with a probable or causal relationship to the LINEA lead which triggered an additional invasive intervention or resulted in patient death
LINEA lead pacing threshold amplitude at 3 months | 3 months after implantation
  Mean ventricular pacing threshold amplitude

SECONDARY OUTCOMES:
Success rate of LINEA lead minimum sensed amplitude | 3 months after implantation
  Proportion of patients with minimum sensed amplitude ≥ 5 mV
General performances of LINEA lead | Implantation, 72 hours from implantation, 1 month, 3 months, 6 months, 18 months, 30 months and 42 months after implantation
  Pacing threshold amplitude, impedance and minimum sensed amplitude obtained with the LINEA lead at each patient's visit. LBB pacing threshold amplitude obtained with the LINEA lead during implantation, as well as the chronaxie measurement
Safety of the LINEA lead | Implantation, 72 hours from implantation, 1 month, 3 months, 6 months, 18 months, 30 months and 42 months after implantation
  LINEA lead complication free rate over time, calculated based on number of Adverse Events and Device Deficiencies related to the lead
Safety of the FLEXIGO delivery catheter and the FLEXIGO slitter | Implantation, 72 hours from implantation, 1 month, 3 months, 6 months, 18 months, 30 months and 42 months after implantation
  FLEXIGO catheter complication free rate, calculated based on number of Adverse Events and Device Deficiencies related to the catheter or the slitter
LINEA lead implantation success rates | Implantation
  Proportion of LINEA leads implanted in the interventricular septum and meeting or not LBBAP criteria
Lead and delivery catheter implantation time | Implantation
  Total procedural time and total fluoroscopic time of each implantation
LINEA lead and FLEXIGO delivery catheter and slitter implantation usability | Implantation
  Handling scores based on a specific questionnaire (scale Very poor/Poor/Acceptable/Good/Very good)
Right Ventricular Autothreshold performances | 3 months after implantation
  - Accuracy - Comparison between the manual ventricular pacing threshold performed by a physician and the in-clinic ventricular pacing threshold provided by the RVAT function at the same pulse width and during the same on-site patient's visit
Evolution of LBBAP capture over time | 18 months after implantation
  - LBBAP capture evolution with analyses of ECGs (i.e. V6 R-wave peak time and V6-V1 interpeak interval) and LBBAP criteria collected

OTHER OUTCOMES:
Early outcome - Absence of Unanticipated Serious Adverse Device Effect (USADE) related to LINEA lead | 1 month after implantation
  Proportion of patients free from USADE. Any event caused by use of the LINEA lead or any accessory packaged with the lead, will be considered as an ADE related to the LINEA lead. The endpoint evaluation will be based on an independent safety events adjudication from a Clinical Events Committee (CEC), based on investigational site reporting
Early outcome - LINEA lead pacing threshold amplitude at 1 month | 1 month after implantation
  Mean ventricular pacing threshold amplitude
Early outcome - Other LINEA lead and FLEXIGO delivery catheter safety and performance | 1 month after implantation
  - Implantation success rate - Proportion of LINEA lead successfully implanted at the interventricular septum and fulfilling or not LBBAP success criteria according to the operator's decision
Early outcome - Other LINEA lead and FLEXIGO delivery catheter safety and performance | 1 month after implantation
  - Short term electrical performances variation - Pacing threshold variation between implantation and 1 month, and electrical performances of the LINEA lead (pacing threshold, impedance and minimum sensed amplitude)
Early outcome - Other LINEA lead and FLEXIGO delivery catheter safety and performance | 1 month after implantation
  - Complication free rate - Proportion of patients free from complication related to the LINEA lead. A complication is defined as a SADE with a probable or causal relationship to the LINEA lead which triggered an additional invasive intervention or resulted in patient death

IPD SHARING:
Plan to Share IPD: No